CLINICAL TRIAL: NCT04859127
Title: Master Student at Kırıkkale University and Physiotherapist
Brief Title: Effects Of Neck Pain Such As Fear Of Movement, Muscle Performance, Disability Etc.
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, BİNNAZ BOZKURT, Master Student (Graduate Student and Researcher), Kırıkkale University
Other Study IDs: kırıkkaleuniversity1.
Record Dates: First submitted 2021-04-13; First posted 2021-04-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: The criteria for inclusion in the study were determined as voluntary patients between the ages of 18-65 with neck pain lasting more than 3 months who were clinically diagnosed with chronic neck pain by a specialist physician.
  Within the scope of the evaluation for the assessment of pain by visual analog scale (VAS), standard evaluation posture Postural Analysis, range of motion for the evaluation of Elektrogonyometer, Nov stabilizer and force evaluation for a hand-held Dynamometer, Nov for brevity, brevity reviews left internal rotator muscles of the pectoral muscles with standard, fear of movement kinezyofobi Tampa scale for the assessment of the neck in apology etc.
  Interventions: Other: effects of neck pain
- Control Group: Asymptomatic individuals between the ages of 18-65 who have not experienced neck pain during the last 1 year will be included in the control group. Within the scope of the evaluation for the assessment of pain by visual analog scale (VAS), standard evaluation posture Postural Analysis, range of motion for the evaluation of Elektrogonyometer, Nov stabilizer and force evaluation for a hand-held Dynamometer, Nov for brevity, brevity reviews left internal rotator muscles of the pectoral muscles with standard, fear of movement kinezyofobi Tampa scale for the assessment of the neck in apology etc.
  Interventions: Other: effects of neck pain

INTERVENTIONS:
Other: effects of neck pain — Within the scope of the evaluation for the assessment of pain by visual analog scale (VAS), standard evaluation posture Postural Analysis, range of motion for the evaluation of Elektrogonyometer, Nov stabilizer and force evaluation for a hand-held Dynamometer, Nov for brevity, brevity reviews left internal rotator muscles of the pectoral muscles with standard, fear of movement kinezyofobi Tampa scale for the assessment of the neck in apology, questioning of the status of the inquiry Neck Disability Survey, stars in the evaluation of balance dynamic balance test, stand on one leg Test in the evaluation of static balance, dynamic balance and physical performance Term rise and walk test, gait speed for the assessment of the 10-meter walk test and dual-task for the evaluation of the motor-the motor and motor-Cognitive dual-task will be used for the evaluation.

SUMMARY:
INTRODUCTION Non-specific chronic neck pain is one of the most common musculoskeletal disorders today. Factors related to neck pain are diverse and can affect the person in different ways. In order to determine the appropriate physical therapy and rehabilitation program for patients, the functional status of the patients should be evaluated carefully and the factors affecting this situation and the relationships between them should be taken into account. Parameters such as pain, balance, disability, muscular performance are associated with neck pain.

The aim of our study is to examine the relationship between pain and kinesophobia and muscle performance, balance and dual task in individuals with nonspecific chronic neck pain and to compare them with asymptomatic individuals.

Materials and Methods:

The study included 44 individuals aged 18-65 who applied to Kırıkkale University Faculty of Medicine Physical Medicine and Rehabilitation Clinic and were diagnosed with non-specific chronic neck pain by a specialist, and 44 asymptomatic individuals between the ages of 18-65 who did not experience neck pain for the last 1 year for the control group. will be. A total of 88 individuals will be included. We will evaluate kinesiophobia, pain density, muscles performance, dual task etc.

FINDINGS AND DISCUSSION: Data acquired at the end of this study will be compared by using appropriate statistical methods and then it will be discussed in comparison with national and international literature.

DETAILED DESCRIPTION:
METHOD DETAIL

1. Pain Severity Assessment Pain assessment is a complex task with a number of goals, including determining the meaning of pain for the patient, understanding the causes as well as consequences of pain, and determining the effectiveness of pain management. The Visual Analogue Scale (VAS) is one of the most widely used measurement methods in pain measurement. GAS is a one-dimensional linear scale. It is easy to use, the results are reproducible, and it can be used in a wide variety of environments. VAS is a continuous scale consisting of a 10 cm (100 mm) horizontal or vertical line. While determining the pain intensity; (0 points) qualifies as "no pain" and (100 points on a 100 mm scale) "pain as bad as possible" or "worst pain imaginable". While calculating the pain severity score, the patient chooses the appropriate point from the 10 cm line. It indicates the presence of no pain on a scale of 100 mm (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), severe pain (75-100 mm).
2. Posture Evaluation The postures of the subjects participating in the study will be evaluated by the standard posture analysis method. Round shoulder, anterior tilt, kyphosis, etc. postural disturbances will be recorded.
3. Joint Range of Motion Assessment (ARA) Normal range of motion will be evaluated using an Electrogoniometer. In the sitting position, the flexion, extension, lateral flexion and rotation movements of the relevant region will be measured and recorded. Evaluations of joint movements will be made in 3 repetitions and the average value of these 3 measurements will be determined by calculating.
4. Muscular Strength Assessment Muscle strength of the neck flexor and extensor muscles will be measured using the Stabilizer (Chattanooga Stabilizer Group Inc., Hixson, TN), and Hand-Held Dynamometer.
5. Assessment of Muscular Endurance Resistance measurements will be made on the extensor and flexor muscles of the neck in a stable position, in the supine and prone positions, respectively. While measuring the endurance of the extensor neck muscles, the patient's legs will be straight and his arms will be positioned around the head. Loads of 2 and 4 kilograms will be applied for women and men, respectively. The test will be done by stretching the head just above the bed and lifting it up for as long (seconds) as possible. Endurance evaluation of the deep cervical flexor muscles will be started with the subject in the hooked position on the back and the hands in the free position on the abdomen. The case will be asked to raise his head slightly high enough for the index and middle finger of a hand to pass along with the instruction. After the patient is taught this position, a slight amount (30%) of craniocervical flexion will be requested from the beginning as if yes. While the subject is in this position, the hand support will be pulled slightly and the test will be started in this position. The time in which the craniocervical maintains the position while maintaining flexion will be recorded in seconds. The test will be terminated when the patient does one of the four situations stated below;

1- In cases where the patient feels a lot of pain and states that he cannot continue 2- In cases where the patient does not feel any pain but endurance ends 3- If the physiotherapist determines that the patient has lost the craniocervical flexion position despite maintaining the position 4- If the physiotherapist observes that the subject lifts his head higher than it should be, the endurance test ends.

The resistance of the case for 60 seconds will be considered sufficient for the termination of the endurance test.

6.Muscular Shortness Assessment In order to determine the muscle shortness of individuals; Standard shortness will be assessed for the pectoral muscles and the adductor and internal rotator muscles.

7. Kinesiophobia Assessment In evaluating the level of kinesiophobia, the 17-question "Tampa Kinesophobia Scale (TSI)" developed by Vlaeyen et al. and validated in Turkish by Tunca Yılmaz and her colleagues will be used. The higher the calculated score, the higher the person's fear of movement will be determined.

8. Spouse Apology Assessment The Neck Disability Index (NDI) is the most widely used tool to measure perceived disability associated with neck pain. The Turkish version of the scale, made by Aslan et al. consists of 10 parts. The questionnaire includes parameters of pain intensity, self-care, lifting, reading, headaches, concentration, work, driving, sleep and activities of daily living. As a result of scoring; (0-4 points) means no disability, (5-14 points) mild disability, (15-24 points) moderate disability, (25-34 points) severe disability and (35 points and above) total disability .

9.Dynamic Balance Assessment

Star Balance Test (YDT) will be used in dynamic balance assessment. Participants stand in the middle of a platform consisting of eight lines that extend at an angle of 45 ° to each other. During the test, the person should rest on one lower limb while reaching as far as possible along each of the eight lines with the other. 8 directions anterior (A), anterolateral (AL), lateral (L), posterolateral (PL), posterior (P), posteromedial (PM), medial (M) and anteromedial (AM). The person is asked to make a light touch on the determined lines and return the reaching leg to the center, and to stand with one leg in the center. Then the maximum distance reached is recorded. If it will be done with the left foot, it is requested to lie counterclockwise, if it will be done with the right foot, it is desired to lie in a clockwise direction. The following formula is used to calculate the star balance test score:

YDT score = (Reaching distance / Leg length) * 100 .

10. Static Balance Evaluation Static balance will be evaluated with the "One Leg Standing Test (TBÜD)". This test measures static balance and static standing ability. It also provides information about the fall risk of the person. The time starts when the person lifts one leg from the ground, and ends when he puts it on the ground. The total time is recorded by the clinician. If the person can keep one leg up for 30 seconds, the test is terminated. If the position can be maintained for less than 10 seconds, the person has an imbalance, and if it is maintained for less than 5 seconds, it can be interpreted that there is a risk of falling for the person.

11. Dynamic Balance and Physical Performance Evaluation The "Timed Get Up and Go Test" will be used for dynamic balance and physical performance evaluation. In this test, the participant should get up without holding the arms of the standard chair in which he or she sits, and after 3 meters of walking, he must return to the chair without touching anything.

12. Walking Speed Assessment The 10 meter walking test will be used to evaluate the walking speed. The person will be asked to walk 14 meters, but the first 2 and the last 2 meters will not be evaluated. It will be calculated in seconds in how long a person takes this distance while walking normally. The time will be recorded in meters / second (m / s), provided that the time starts when the person's foot is at the starting line of the 2nd meter and ends when the 12 meter line is crossed.

13. Dual-Task Assessment The dual task will be evaluated motor-motor and motor-cognitively during walking. Participants will be subjected to 6 different walks. Participants will be given a clear explanation about the tests before the tests and will be informed about their comfort. Participants will be given a trial test only once before the test.

* 10 m Walking Test (single duty)
* 10 m Walking Test + The task of carrying 2 glasses of water on a standard tray without spilling the water in the glass (motor-motor dual duty)
* 10 m Walking Test + A task of counting 6 from any two-digit number selected by the clinician during the test (motor-cognitive dual task)
* Timed Get Up and Go Test (single task)
* Timed Get Up and Go Test + The task of carrying 2 glasses of water on a standard tray without spilling the water in the glass (motor-motor dual duty)
* Timed Get Up and Go Test + The task of counting 6 from any two-digit number selected by the clinician during the test (motor-cognitive dual task)

During the tests, single tasks will be included for reference. The completion times of the motor-motor and motor-cognitive dual tasks, which are evaluated 2 in 2 each with 4 different walking forms, will be recorded and the result will be reached. The following calculation method will be used for the result:

Dual Mission Effect = (Single Mission Performance - Dual Mission Performance) / Single Mission Performance x 100

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria in the Study;

1. Between the ages of 18-65,
2. Have neck pain that lasts longer than 3 months,
3. Volunteer patients diagnosed with chronic neck pain by a specialist,

Inclusion criteria in the control group;

1. Has not experienced neck pain for the last 1 year,
2. Asymptomatic individuals between the ages of 18-65,

Exclusion Criteria:

The criteria for exclusion from the study;

1. Having had cervical spine and shoulder surgery,
2. Neck pain caused by different pathologies (tumor, rheumatoid arthritis, ankylosing spondylitis, fracture, dislocation),
3. With cord compression and findings (L'hermitte sign is positive),
4. Having severe radiculopathy (Upper limb tension tests are positive),
5. Have osteoporosis,
6. It has been identified as having shoulder pain and any shoulder pathology (Rotator Cuff tear, shoulder impingement syndrome, etc.).

Exclusion criteria for the control group; 1. Those who have experienced neck pain in the last 1 year, 2. Different pathologies (inflammatory diseases, neoplasia, vertebral dislocation fracture history) 3. Previous cervical spine and shoulder surgery, 4. Those with advanced osteoporosis causing compression fracture, 5. Those with shoulder pathology,

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Between the ages of 18-65 men and women.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Investigation Of The Relationship Between Pain And Fear Of Motion And Muscle Performance, Balance And Dual Task In Individuals With Non-Specific Chronic Neck Pain And Comparing With Asymptomatic Individuals | 16 weeks
  Pain Intensity Assessment VAS out of 10 points ROM Evaluation Electrogoniometer the measured angle Muscle Strength Assessment will be measured the neck flexor and extensor muscles, Stabilizer and Hand-Held Dynamometer and recorded in newtons and mm / hg Muscular Endurance Assessment the extensor and flexor muscles of the neck will be recorded (s) Muscle Shortness Assessment pectoral, adductor and internal rotator muscles (short-normal-long) Kinesiophobia Assessment Tampa Kinesophobia Scale (score) Neck Disability Assessment Neck Disability Index (score) Dynamic Balance Assessment Star Balance Test (cm) SBT score = (Reaching distance / Leg length) * 100 Static Balance Assessment One-Standing Standing Test (s) Physical PerformanceTUG Test (s) Walking Speed Assessment 10 m walking test (s) Dual Task Assessment motor-motor and motor-cognitive during walking (s) Dual Task Effect = (Single Task - Dual Task ) / Single Task x 100 (s=seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale Üniversitesi, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We dont decide yet